CLINICAL TRIAL: NCT00450788
Title: The Golestan Cohort Study of Esophageal Cancer
Brief Title: Esophageal Cancer in Northeastern Iran
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907120; 07-C-N120
Record Dates: First submitted 2007-03-17; First posted 2007-03-22 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2025-07-11

CONDITIONS: Esophageal Cancer; GI Disease
Keywords: Etiology; Carcinogens; Esophageal Cancer; Natural History
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Golestan Cohort: Cohort of adults from Golestan region in Iran

SUMMARY:
Background:

-Esophageal cancer is the most common cancer in Iran s Golestan Province. Nutritional deficiencies, ethnicity and environmental exposures might contribute to the development of this disease.

Objectives:

-To better understand the cause of esophageal cancer in Golestan Province and to reduce its occurrence there.

Eligibility:

-Adults from the Gonbad, Aq-Qala and Kalaleh districts of eastern Golestan Province in Iran.

Design:

* The study is a collaboration between NIH, the Digestive Disease Research Center of Teheran University of Medical Sciences, and the International Agency for Research on Cancer.
* Participants complete a lifestyle questionnaire and food frequency questionnaire.
* Samples of participants blood, urine, hair and toenail clippings are obtained.

DETAILED DESCRIPTION:
Esophageal cancer is the sixth most common cause of cancer death worldwide, killing over 380,000 people each year. Over 80% of esophageal cancers occur in developing countries, where the great majority of cases are squamous cell carcinomas. Esophageal cancer is characterized by striking geographic variation in incidence. One remarkable high-risk area, called the Central Asian Esophageal Cancer Belt, stretches from the Caspian Sea across Central Asia to northern China and includes focal areas with recorded incidence rates greater than 100/10s/year in both genders. For the past 20 years, D CEG investigators have studied esophageal and gastric cancer in one of these extremely high-risk areas, Linxian, China, at the eastern end of the Belt. While these studies have discovered new risk factors for esophageal cancer in this region, they have produced an incomplete explanation of the etiology of this disease. Now we have the opportunity to perform similar studies in another of these extremely high-risk areas, Golestan Province, Iran, at the other end of the high-risk Belt. The people of Golestan, in northeastern Iran, are geographically, culturally and ethnically quite different from the people of Linxian, and they appear to be similar only in their extraordinarily high rates of esophageal cancer. Performing similar studies in these two exceptional populations will give us a better chance to identify important new modifiable risk factors for esophageal cancer in both places.

Our cohort study is a collaboration between the Digestive Disease Research Center of Tehran University of Medical Sciences (DDRC), the International Agency for Research on Cancer (IARC), and DCEG. The study has recruited 50,000 adults in three administrative districts of eastern Golestan Province. Baseline assessments included lifestyle questionnaire, a semi-quantitative food frequency questionnaire, and collection of blood, hair, nails and urine. Follow up will includes active surveillance by a study team, aided by a comprehensive health network in the rural areas, a GI referral clinic in the largest town, and a provincial cancer registry. The main hypotheses include dietary hypotheses (low consumption of fruits and vegetables, high consumption of hot tea), exposure to potential carcinogens (tobacco, PAHs from non-tobacco sources), novel exposures (opium, animal contact), and genetic susceptibility. Some cross sectional and a few total mortality analyses have been completed. Annual follow-up is ongoing.

ELIGIBILITY:
* Ages 40 to 75

  * Patients with esophogeal cancer

Ages: 30 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study has recruited 50,000 adults in three administrative districts of eastern Golestan Province. Baseline assessments included lifestyle questionnaire, a semi-quantitative food frequency questionnaire, and collection of blood, hair, nails and urine. Follow up will includes active surveillance by a study team, aided by a comprehensive health network in the rural areas, a GI referral clinic in the largest town, and a provincial cancer registry.
Sampling Method: Probability Sample
Enrollment: 50045 (Actual)
Dates: Start 2007-03-15

PRIMARY OUTCOMES:
cancer incidence | continuous
  The main hypotheses include dietary hypotheses (low consumption of fruits and vegetables, high consumption of hot tea), exposure to potential carcinogens (tobacco, PAHs from non-tobacco sources), novel exposures (opium, animal contact), and genetic susceptibility.

SECONDARY OUTCOMES:
Mortality | Continuous
  Some cross sectional and a few total mortality analyses have been completed.

CONTACTS AND LOCATIONS:
Overall Officials: Christian C Abnet, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Digestive Disease Research Institute, Tehran, Iran

REFERENCES:
- [Background] Pourshams A, Khademi H, Malekshah AF, Islami F, Nouraei M, Sadjadi AR, Jafari E, Rakhshani N, Salahi R, Semnani S, Kamangar F, Abnet CC, Ponder B, Day N, Dawsey SM, Boffetta P, Malekzadeh R. Cohort Profile: The Golestan Cohort Study--a prospective study of oesophageal cancer in northern Iran. Int J Epidemiol. 2010 Feb;39(1):52-9. doi: 10.1093/ije/dyp161. Epub 2009 Mar 30. No abstract available. PMID 19332502
- [Background] Malekshah AF, Kimiagar M, Saadatian-Elahi M, Pourshams A, Nouraie M, Goglani G, Hoshiarrad A, Sadatsafavi M, Golestan B, Yoonesi A, Rakhshani N, Fahimi S, Nasrollahzadeh D, Salahi R, Ghafarpour A, Semnani S, Steghens JP, Abnet CC, Kamangar F, Dawsey SM, Brennan P, Boffetta P, Malekzadeh R. Validity and reliability of a new food frequency questionnaire compared to 24 h recalls and biochemical measurements: pilot phase of Golestan cohort study of esophageal cancer. Eur J Clin Nutr. 2006 Aug;60(8):971-7. doi: 10.1038/sj.ejcn.1602407. Epub 2006 Feb 8. PMID 16465196
- [Background] Pourshams A, Saadatian-Elahi M, Nouraie M, Malekshah AF, Rakhshani N, Salahi R, Yoonessi A, Semnani S, Islami F, Sotoudeh M, Fahimi S, Sadjadi AR, Nasrollahzadeh D, Aghcheli K, Kamangar F, Abnet CC, Saidi F, Sewram V, Strickland PT, Dawsey SM, Brennan P, Boffetta P, Malekzadeh R. Golestan cohort study of oesophageal cancer: feasibility and first results. Br J Cancer. 2005 Jan 17;92(1):176-81. doi: 10.1038/sj.bjc.6602249. PMID 15597107